CLINICAL TRIAL: NCT04049994
Title: Immunomodulation Therapy for Primary Prevention of Urinary Tract Infections in Patients With Spinal Cord Injury During First Rehabilitation: a Randomized Controlled Pilot Study
Brief Title: Immunomodulation Therapy for Urinary Tract Infections
Acronym: UROVAXOM-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Swiss Spinal Cord Injury Cohort Study (SwiSCI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-22
Record Dates: First submitted 2019-07-10; First posted 2019-08-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries; Urinary Tract Infections
Keywords: spinal cord injury; neurogenic lower urinary tract dysfunction; urinary tract infection; immunotherapy; immunomodulation; immunostimulation; E. coli; Uro-Vaxom
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunomodulation (Experimental): Lyophilized lysate of 18 E. coli strains (6 mg) for oral application. A treatment lasts 90 days (one capsule daily).
  Interventions: Drug: Uro-Vaxom
- Placebo (Placebo Comparator): Oral placebo tablet once daily for 90 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Uro-Vaxom — Uro-Vaxom® (OM Pharma SA, Meyrin, Switzerland) is a lyophilized lysate of 18 E. coli strains.
  Arms: Immunomodulation
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: Placebo

SUMMARY:
Urinary tract infections (UTI) represent one of the most common morbidities in individuals with spinal cord injury (SCI) and reason for re-hospitalization. The consequences of recurrent UTI are a decrease in quality of life and considerable health costs. Immunomodulation therapy with UroVaxom is a very promising method for the prevention of UTI, however data in individuals with SCI are very limited. The primary objective of this pilot study is to evaluate the feasibility (recruitment rate, patient attrition, compliance, assessment procedures etc.) of a main trial. A secondary objective is to collect data for an informed sample size calculation. Furthermore, the clinical and biological changes after immunomodulation therapy will be investigated.

This is a randomized, placebo-controlled, mono-centric pilot study investigating the feasibility of a main trial regarding the effectiveness of immunomodulation with UroVaxom in the prevention of UTI and the effect on the immune system in individuals with acute SCI during primary rehabilitation. There will be two parallel groups of 12 participants each. Group allocation will be based on a block-randomization stratified according to sex. Study participants and outcome assessors will be blinded to the group allocation. The nursing staff will be unblinded and will administer the treatment and the placebo. Study participants will either receive Uro-Vaxom (one tablet / day) or an off-the-shelf placebo for 90 days. After termination of the treatment, the study participants will be followed for 12 months. Blood and urine samples will be taken before and 90 days, 6 months and 12 months after treatment start.

ELIGIBILITY:
Inclusion Criteria:

* acute SCI (within 8 weeks after SCI)
* onset of SCI within 72h
* age from 18 to 70 years
* informed consent as documented by signature

Exclusion Criteria:

* known hypersensitivity to investigational product,
* other immunomodulation therapy,
* immunosuppressant therapy,
* oncological condition or therapy,
* autoimmune diseases, nephropathy, bladder stones,
* women who are pregnant (pregnancy test) or breast feeding,
* participation in another study with an investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
randomization rate | at study completion, an average of 2 years
  proportion of eligible patients who were enrolled

SECONDARY OUTCOMES:
positive screening rate | at study completion, an average of 2 years
  proportion of eligible patients who were screened
retention rate | at study completion, an average of 2 years
  treatment-specific retention rate
drop-out rate | at study completion, an average of 2 years
  rate of enrolled study participants who do not complete the study protocol
urine culture result | during follow-up of 12 months
  bacteria species isolated from urine of study participants
change in urinary immunoglobulin A levels | time 0 and 12 months
  concentration (mg/dl) of immunoglobulin A in the urine
count of urinary tract infection | during follow-up of 12 months
  occurrence of a symptomatic urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, Prof. Dr., Principal Investigator — Swiss Paraplegic Centre
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valido E, Bertolo A, Wollner J, Pannek J, Krebs J, Stoyanov J. Effects of Uro-Vaxom vs. placebo on the urinary tract microbiome in individuals with spinal cord injury in a randomized controlled pilot trial (Uro-Vaxom pilot). Sci Rep. 2025 Apr 14;15(1):12825. doi: 10.1038/s41598-025-96939-y. PMID 40229352
- [Derived] Krebs J, Stoyanov J, Wollner J, Valido E, Pannek J. Immunomodulation for primary prevention of urinary tract infections in patients with spinal cord injury during primary rehabilitation: protocol for a randomized placebo-controlled pilot trial (UROVAXOM-pilot). Trials. 2021 Oct 4;22(1):677. doi: 10.1186/s13063-021-05630-w. PMID 34607600